CLINICAL TRIAL: NCT00071435
Title: Movement Related Cortical Potentials in Primary Lateral Sclerosis
Brief Title: Brain Function in Primary Lateral Sclerosis
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040017; 04-N-0017
Record Dates: First submitted 2003-10-22; First posted 2003-10-23 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-02

CONDITIONS: Motor Neuron Disease
Keywords: EEG; Voluntary Movement; Motor Cortex; Reaction Time; Corticospinal; Primary Lateral Sclerosis; PLS; Healthy Volunteer; HV
MeSH Terms: conditions — Motor Neuron Disease

SUMMARY:
This study will examine whether the motor cortex (the part of the brain that controls movement) works properly in patients with primary lateral sclerosis (PLS), a disorder in which voluntary movements are very slow.

Healthy volunteers between 40 and 75 years of age and patients with ascending PLS (a subset of PLS) may be eligible for this study. Patients with ascending PLS have a slowing of finger-tapping movements that corresponds to a particular abnormality of certain neuronal (nerve cell) activity.

Participants perform a finger-tapping reaction time exercise while brain wave activity (electroencephalography, or EEG) and muscle activity (electroymogram, or EMG) are measured. The subject is seated in front of a computer screen. A signal appears on the screen and the subject taps a key as quickly as possible in response to the signal.

For the EEG, brain activity is recorded by placing electrodes (small metal discs) on the scalp with an electrode cap or glue-like substance. A conductive gel is used to fill the space between the electrodes and the scalp to make sure there is good contact between them. The brain waves are recorded while the subject taps his or her fingers very slowly. For the surface EMG, electrodes filled with a conductive gel are taped to the skin.

Participants also undergo magnetic resonance imaging (MRI). This test uses a strong magnetic field and radio waves to obtain images of the brain. During the procedure, the subject lies still on a table that can slide in and out of the scanner - a narrow metal cylinder. Scanning time varies from 20 minutes to 3 hours, with most scans lasting between 45 and 90 minutes. Subjects can communicate with the MRI staff at all times during the scan and can ask to be moved out of the machine at any time.

DETAILED DESCRIPTION:
Objective: Primary Lateral Sclerosis (PLS) is a clinical syndrome of progressive spasticity. Patients with PLS have slow voluntary movements. In PLS, degeneration of corticospinal tracts disrupts the communication between the motor cortex and motor neurons. Normally, voluntary movements are preceded by EEG waveform changes that begin before the movement occurs. These waveforms are called movement related cortical potentials (MRCPs). The first part of the MRCP represents neural activity in the motor cortex. The goal of this study is to determine whether the motor cortex and pre-motor cortex operate normally to generate these intrinsic signals for voluntary movement in patients with PLS.

Study population: Patients with PLS of at least 3 years duration with slow finger tapping movements will be studied. Patients must fulfill the clinical criteria for the ascending subtype of PLS. They must also have a loss of corticospinal excitability as measured by transcranial magnetic stimulation. Age matched normal volunteers will be studied as a control group.

Design: Patients and normal volunteers will undergo a session of EEG recording while making slow finger tapping movements. They will have an MRI of the brain, for the purpose of localizing dipole positions of the MRCP components.

Outcome parameters: The peak amplitudes of components of the MRCPs will be compared between patients and a healthy control group as the primary outcome measure. Localization of the dipoles of the components is a secondary outcome measure.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients

1. Ages 40-75
2. Fulfill the proposed diagnostic criteria for PLS of Pringle 1992.
3. Have an ascending course of symptom progression.
4. Slow hand movements, as determined by measuring finger-tapping speeds of 20-65 taps in 15 s.
5. Absent motor evoked potentials in hand muscles with 100% output of the MagStim200 transcranial magnetic stimulator.

Normal Volunteers

Healthy adult volunteers ages 40-75 who are willing to participate.

EXCLUSION CRITERIA:

1. Neurological diseases or conditions other than PLS.
2. Implanted devices, such as pumps, pacemakers, or metal fragments in the skull or eye.
3. Pregnancy as determined by urine pregnancy test within 48 hours of MRI study in women of childbearing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36
Dates: Start 2003-10; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Rowland LP. Primary lateral sclerosis: disease, syndrome, both or neither? J Neurol Sci. 1999 Nov 15;170(1):1-4. doi: 10.1016/s0022-510x(99)00183-5. No abstract available. PMID 10540028
- [Background] Swash M, Desai J, Misra VP. What is primary lateral sclerosis? J Neurol Sci. 1999 Nov 15;170(1):5-10. doi: 10.1016/s0022-510x(99)00184-7. PMID 10540029
- [Background] Sasaki S, Iwata M. Ultrastructural study of Betz cells in the primary motor cortex of the human brain. J Anat. 2001 Dec;199(Pt 6):699-708. doi: 10.1046/j.1469-7580.2001.19960699.x. PMID 11787823